CLINICAL TRIAL: NCT04424485
Title: Near-infrared (NIR) Fluorescence Imaging With Indocyanine Green (ICG) for Identification of Sentinel Lymph Nodes and Parathyroid Glands During Total Thyroidectomy: Prospective Randomized Clinical Trial
Brief Title: Near-infrared Fluorescence With Indocyanine Green for Identification of Sentinels and Parathyroids During Thyroidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ethem Unal, M.D., PhD, Associate Prof of Surgery & Surgic, A. Prof. of General Surgery and Surgical Oncology, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: B.10.1.TKH.4.34.H.GP.0.01/213
Record Dates: First submitted 2020-06-02; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Thyroid Cancer; Thyroid Carcinoma, Papillary; Thyroid Metastases; Thyroid Neoplasms; Sentinel Lymph Node; Lymph Node Metastases
Keywords: Near-infrared (NIR) fluorescence; Total thyroidectomy; Parathyroid glands; Indocyanine green (ICG); Central lymph node dissection
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary; Lymphatic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thyroid carcinoma patients (biopsy-proven)-Total thyroidectomy (Active Comparator): Control group-Total thyroidectomy (TT) with central lymph node dissection (CLND) procedure for patients with papillary thyroid carcinoma (PTC)
  Standard TT+CLND procedure only
  Interventions: Procedure: Total thyroidectomy (TT); Procedure: Central lymph node dissection (CLND)
- Thyroid carcinoma patients (biopsy-proven)-Sentinel lymph node (Experimental): Experimental group- Sentinel lymph node dissection (SLND) after intratumoral indocyanine green (ICG) injection and visualization of all 4 parathyroid glands with infra-red (NIR) fluorescence after intravenous (iv) ICG injection, during total thyroidectomy and central lymph node dissection (CLND).
  TT+CLND with NIR fluorescence ICG
  Interventions: Procedure: Total thyroidectomy (TT); Procedure: Central lymph node dissection (CLND); Diagnostic Test: Sentinel lymph node (SLN) bopsy; Diagnostic Test: Identification of parathyroid glands (PGs)

INTERVENTIONS:
Procedure: Total thyroidectomy (TT) — Standard TT procedure for thyroid carcinoma, for both groups
Procedure: Central lymph node dissection (CLND) — Standard CLND for thyroid carcinoma, for both groups
Diagnostic Test: Sentinel lymph node (SLN) bopsy — Intrathyroidal injection of ICG for SL biopsy, for only experimental group
  Arms: Thyroid carcinoma patients (biopsy-proven)-Sentinel lymph node
Diagnostic Test: Identification of parathyroid glands (PGs) — Near-infrared (NIR) fluorescence visualization of PGs, for only experimental group
  Arms: Thyroid carcinoma patients (biopsy-proven)-Sentinel lymph node

SUMMARY:
Indocyanine green (ICG) is a water-soluble organic dye that is cleared totally through the hepatobiliary system. It has a half-life of 3-4 mins, which allows repeated applications. Near-infrared (NIR) fluorescence imaging with indocyanine green (ICG) imaging has been recently introduced, and has been suggested as a useful tool for the identification and preservation of the parathyroid glands (PGs) during total thyroidectomy (TT). ICG can also be used for sentinel lymph node (SLN) biopsy to predict the micrometastases in central lymph nodes (CLN) in thyroid carcinoma, and central lymph node dissection can reduce local recurrence.

DETAILED DESCRIPTION:
Incidence of thyroid cancer has doubled between 1980 and 2020, and it is now the fifth most common malignant tumor among women. The majority are papillary thyroid cancer (PTC), and TT is the procedure of choice. Since the micrometastasis rate of the central lymph nodes (CLNs) is about 30% to 90% in PTC, CLN dissection can improve the prognosis and reduce tumor recurrence as well as provide accurate information for the evaluation of tumor staging. However, TT procedure has some important complications such as vocal cord paralysis (VCP) and hypocalcemia (due to accicental parathyroidectomy or damage to the parathyroid gland-PG- vasculature). Use of intraoperative nerve monitoring (IONM) has reduced the rate of VCP. However, the incidence of postoperative hypocalcemia is still high (15-70%), and it is now the most common complication of TT. Intraoperative identification of SLNs and PGs can help surgeon to overcome these problems.

ELIGIBILITY:
Inclusion Criteria:

* Thyroid carcinoma patients (biopsy/cytology-proven) suitable for total thyroidectomy procedure
* Patients at or over 17 years

Exclusion Criteria:

* Previous thyroid surgery
* Patients below 17 years

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Involvement of sentinel lymph node (presence/absence of tumor cell: positive or negative) by histopathological examinatiion | 1 year
  Intrathyroidal injection of indocyanine green (ICG) dye to identify sentinel lymph node (SLN) for biopsy
Identification of parathyroid glands (PGs) by NIR/ICG camera detected high-contrast | 1 year
  İntravenous injection of ICG dye, to identify PGs under NIR (High-contrast fluorescence seen or not)

SECONDARY OUTCOMES:
Central lymph node dissetion (CLND) | 1 year
  Number of positive lymph nodes (micrometastases)

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Education and Research Hospital, Department of General Surgery, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Excel data is available upon request at drethemunal@gmail.com
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year
Access Criteria: Please request study protocol and data (when available) at drethemunal@gmail.com

REFERENCES:
- [Result] Zhang X, Shen YP, Li JG, Chen G. Clinical feasibility of imaging with indocyanine green combined with carbon nanoparticles for sentinel lymph node identification in papillary thyroid microcarcinoma. Medicine (Baltimore). 2019 Sep;98(36):e16935. doi: 10.1097/MD.0000000000016935. PMID 31490376
- [Result] Spartalis E, Ntokos G, Georgiou K, Zografos G, Tsourouflis G, Dimitroulis D, Nikiteas NI. Intraoperative Indocyanine Green (ICG) Angiography for the Identification of the Parathyroid Glands: Current Evidence and Future Perspectives. In Vivo. 2020 Jan-Feb;34(1):23-32. doi: 10.21873/invivo.11741. PMID 31882459
- See also: Ethem Unal — https://scholar.google.com.tr/citations?user=6bFlCZwAAAAJ&hl=tr